CLINICAL TRIAL: NCT02153996
Title: Longitudinal Analysis of Plasmodium Falciparum-Specific Immunity in Travelers and Immigrants From Malaria Endemic Areas to the United States
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140121; 14-I-0121
Record Dates: First submitted 2014-05-31; First posted 2014-06-03 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-03-15

CONDITIONS: Malaria
Keywords: Malaria Immunity Longevity
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Plasmodium falciparum malaria is a major cause of morbidity and mortality in tropical and sub-tropical areas worldwide. Repeated P. falciparum infections in endemic areas induce protective immunity, thus providing optimism that an effective malaria vaccine can be developed. Key to the development of such a vaccine is an understanding of the immune mechanisms underlying protection and the longevity of these responses in the absence of continuous P. falciparum exposure. Anecdotal evidence suggests clinical immunity to malaria wanes within months to years after an immune individual leaves an endemic area. A detailed, systematic description of the quality and longevity of the P. falciparum-specific humoral and cellular immune responses in such individuals over time in the absence of ongoing exposure is lacking.

This protocol will attempt to fill this knowledge gap through comprehensive longitudinal immunological analyses of two populations of healthy adult volunteers: 1) naive travelers returning from malaria endemic areas recently treated (within 2 weeks) for acute P. falciparum malaria and referred from hospitals in the metropolitan Washington DC area; and 2) immigrants from malaria endemic areas living in the metropolitan Washington DC area with serologic evidence of past P. falciparum exposure. In both groups, venipuncture and possibly apheresis will be performed for the isolation of plasma, RNA and peripheral blood mononuclear cells (PBMCs) which will be analysed to understand the components of innate and adaptive immunity to malaria. Na(SqrRoot) ve travelers returning from malaria endemic areas recently treated for acute malaria will undergo venipuncture at enrollment, then once every 2 weeks for 2 months, then every 3 months for 1 year, and then every 6 months for up to 5 years. Immigrants will be seen every three months for one year and then every six months for up to 5 years. All subjects who return to the U.S. from a malaria endemic area will be evaluated within two weeks of return for repeat venipuncture and will restart the same sequence of blood draws as naive travelers. Optional apheresis will be performed on both na(SqrRoot) ve travelers and immigrants at enrollment, at 1, 6, and 12 months, then yearly therafter.

The primary objective is to estimate the quality and longevity of P. falciparum-specific humoral and cellular immune responses in the absence of ongoing P. falciparum exposure in both returned na(SqrRoot) ve travelers and immigrants. The secondary objective is to compare the P. falciparum-specific humoral and cellular immune response in na(SqrRoot) ve travelers and immigrants to individuals in malaria-endemic areas enrolled in ongoing LIG protocols in Mali.

...

DETAILED DESCRIPTION:
Plasmodium falciparum malaria is a major cause of morbidity and mortality in tropical and sub-tropical areas worldwide. Repeated P. falciparum infections in endemic areas induce protective immunity, thus providing optimism that an effective malaria vaccine can be developed. Key to the development of such a vaccine is an understanding of the immune mechanisms underlying protection and the longevity of these responses in the absence of continuous P. falciparum exposure. Anecdotal evidence suggests clinical immunity to malaria wanes within months to years after an immune individual leaves an endemic area. A detailed, systematic description of the quality and longevity of the P. falciparum-specific humoral and cellular immune responses in such individuals over time in the absence of ongoing exposure is lacking.

This protocol will attempt to fill this knowledge gap through comprehensive longitudinal immunological analyses of two populations of healthy adult volunteers: 1) naive travelers returning from malaria endemic areas recently treated (within 2 weeks) for acute P. falciparum malaria and referred from hospitals in the metropolitan Washington DC area; and 2) immigrants from malaria endemic areas living in the metropolitan Washington DC area with serologic evidence of past P. falciparum exposure. In both groups, venipuncture and possibly apheresis will be performed for the isolation of plasma, RNA and peripheral blood mononuclear cells (PBMCs) which will be analysed to understand the components of innate and adaptive immunity to malaria. Na(SqrRoot) ve travelers returning from malaria endemic areas recently treated for acute malaria will undergo venipuncture at enrollment, then once every 2 weeks for 2 months, then every 3 months for 1 year, and then every 6 months for up to 5 years. Immigrants will be seen every three months for one year and then every six months for up to 5 years. All subjects who return to the U.S. from a malaria endemic area will be evaluated within two weeks of return for repeat venipuncture and will restart the same sequence of blood draws as naive travelers. Optional apheresis will be performed on both na(SqrRoot) ve travelers and immigrants at enrollment, at 1, 6, and 12 months, then yearly therafter.

The primary objective is to estimate the quality and longevity of P. falciparum-specific humoral and cellular immune responses in the absence of ongoing P. falciparum exposure in both returned na(SqrRoot) ve travelers and immigrants. The secondary objective is to compare the P. falciparum-specific humoral and cellular immune response in na(SqrRoot) ve travelers and immigrants to individuals in malaria-endemic areas enrolled in ongoing LIG protocols in Mali.

ELIGIBILITY:
* INCLUSION CRITERIA:
* All Subjects: Age 18-65
* Agree to have blood specimens stored for future research and genetic studies

Malaria endemicity will be defined according to CDC Yellow Book criteria available at:

http://wwwnc.cdc.gov/travel/yellowbook/2014/chapter-3-infectious-diseases-related-totravel/malaria#3929

NaIve travelers returning from malaria endemic areas recently treated for malaria:

-Treated for acute P. falciparum malaria within 4 weeks of enrolling in this study as determined by clinical and microbiologic evidence (including blood smear) of infection as indicated by medical records

Immigrants from malaria endemic areas:

* Confirmation of having lived in a malaria endemic area through documentation or verifiable detailed immigration history.
* Evidence of past P. falciparum exposure with positive AMA -1 ELISA.

SUBJECT EXCLUSION CRITERIA:

* History of HIV and/or hepatitis C.
* Inadequate peripheral venous access
* Current use of the steroid equivalent of prednisone 20mg/day or more or other systemic immunosuppressants
* Underlying heart disease, lung disease, bleeding disorder, or other conditions that, in the judgment of the investigator, contraindicates study participation
* Temperature greater than or equal to 37.5 (Infinite)C or other clinical evidence of an acute infection
* Currently pregnant (positive urine beta-HCG) or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-05-15; Primary Completion 2016-03-15 (Actual); Study Completion 2016-03-15 (Actual)

PRIMARY OUTCOMES:
Estimate the quality and longevity of P. falciparum-specific humoral and cellular immune responses in the absence of ongoing P. falciparum exposure. | Five years

SECONDARY OUTCOMES:
Compare the P. falciparum-specific humoral and cellular immune response in na(SqrRoot) ve travelers and immigrants to age and sex matched individuals in malaria-endemic areas enrolled in ongoing LIG protocols in Mali. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eugene W Liu, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Trape JF, Rogier C, Konate L, Diagne N, Bouganali H, Canque B, Legros F, Badji A, Ndiaye G, Ndiaye P, et al. The Dielmo project: a longitudinal study of natural malaria infection and the mechanisms of protective immunity in a community living in a holoendemic area of Senegal. Am J Trop Med Hyg. 1994 Aug;51(2):123-37. doi: 10.4269/ajtmh.1994.51.123. PMID 8074247
- [Background] Perignon JL, Druilhe P. Immune mechanisms underlying the premunition against Plasmodium falciparum malaria. Mem Inst Oswaldo Cruz. 1994;89 Suppl 2:51-3. doi: 10.1590/s0074-02761994000600013. PMID 7565132
- [Background] Deloron P, Chougnet C. Is immunity to malaria really short-lived? Parasitol Today. 1992 Nov;8(11):375-8. doi: 10.1016/0169-4758(92)90174-z. PMID 15463545